CLINICAL TRIAL: NCT06226779
Title: Mindful Exercise Baduanjin Versus Brisk Walking for Cognitive Function in Patients With Schizophrenia
Brief Title: Baduanjin Versus Brisk Walking for Cognition in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chen Chyi-Rong, Occupational therapist, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202400006B0
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Exercise; Condition
Keywords: schizophrenia, mindful exercise, exercise, cognition
MeSH Terms: conditions — Schizophrenia; Motor Activity; Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baduanjin (Experimental): Parcipants will practice baduanjin exercise.
  Interventions: Behavioral: Baduanjin exercsie
- Brisk walking (Active Comparator): Parcipants will perform brisk walking activities.
  Interventions: Behavioral: Brisk walking
- health education (Other): Parcipants will receive health education classes and watch sport related videos.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Baduanjin exercsie — The Baduanjin exercise consists of 8 postures, with emphasis on different body parts. The exercise is commonly practiced as follows: (1) 2 hands holding up the heavens, (2) drawing the bow to shoot the eagle, (3) separating the heaven and earth, (4) wise owl gazing backwards, (5) swaying the head and shaking the tail, (6) 2 hands holding the feet to strengthen the waist, (7) clenching the fists and glaring fiercely, and (8) bouncing on the toes.
  Other Names: Mindful baduanjin
  Arms: Baduanjin
Behavioral: Brisk walking — The brisk walking will be gradually increased physical exertion from light to moderate of intensity. During the training period, the heart rate of participants will be monitored.
  Other Names: aerobic walking
  Arms: Brisk walking
Behavioral: Health education — Health education will include lecture classes. Video watching will watch videos which were not aim at improving physical exertion, such as sports games or sports related variety shows
  Other Names: video watching
  Arms: health education

SUMMARY:
The current study intends to recruit participants with schizophrenia for the practice of Baduanjin, brisk walking, and health education after enrollment. The study also including a maintenance program. Cognitive and physical function assessments will be conducted before, after, and during follow-up tests. The research hypothesis posits that both Baduanjin and brisk walking will confer beneficial effects on various aspects of cognitive and physical functions.

DETAILED DESCRIPTION:
Cognitive function deficits are core features in patients with schizophrenia. These deficits need active intervention to prevent functional decline. Baduanjin and brisk walking show promise as interventions in patients with schizophrenia. This study investigated the effects of Baduanjin exercise versus brisk walking in patients with schizophrenia.

This study will be a single-blind, 3-arm, parallel, randomized controlled trial.

A total of 72 patients with schizophrenia will be enrolled and randomly assigned to the Baduanjin group, brisk walking group or control group. The intervention group will practice Badunjin exercise. While participants in brisk walking group will receive brisk walking at the same duration. The controls will watch videos that are not aimed at improving physical exertion. Maintenance programs will also be conducted for participants to encourage practicing in exercise after intervention. All group will undergo evaluation at three time points: baseline, immediately after intervention and 4-week follow up after intervention. The primary outcome will be cognitive function and physical function. Secondary outcomes will include mood, sleep quality, and quality of live.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of schizophrenia according to the DSM-5.
2. Who will be above 20-65 years of age .
3. Having a stable mental status without shift in medication and keep in same dose for at least one month.
4. Being able to walk independently for 50 meters.

Exclusion Criteria:

1. Serious physical conditions that will impede participation, such as cardiovascular disease, musculoskeletal disease or pulmonary system disease.
2. Visual or auditory impairment that precludes completion of assessment.
3. Acute psychosis requiring hospitalization.
4. Presence of severe withdrawal or profound cognitive disability that cause difficulties in following instructions.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity.
Enrollment: 63 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change score of the Brief Assessment of Cognition in Schizophrenia (BACS) | Baseline, immediate after treatment, 4-week follow up
  BACS is a battery of cognition tests that measure verbal memory, working memory, motor speed, verbal fluency, attention and processing speed, and executive function.The BACS is comprised of seven subtests: (1) the List Learning Test, (2) Digit Sequencing Test, (3) Token Motor Test, (4) Category Instance Test, (5) Controlled Oral Word Association Test, (6) Symbol Coding, and (7) Tower of London Test.
Change scores of 6-minute walk test | Baseline, immediate after treatment, 4-week follow up
  This test evaluates cardiovascular fitness and walking speed.
Change scores of 30-second chair stand test | Baseline, immediate after treatment, 4-week follow up
  This test evaluates muscular endurance of lower-extremities.
Change scores of Timed up-and-go test | Baseline, immediate after treatment, 4-week follow up
  This test evaluates functional mobility, agility and balance
Change scores of dual task Timed up-and-go test (manual) | Baseline, immediate after treatment, 4-week follow up
  This test requires carry a cup of water 3 cm from the top of the cup while performing the Timed up-and-go test. It evaluates dual task performance.
Change scores of dual task Timed up-and-go test (cognitive) | Baseline, immediate after treatment, 4-week follow up
  This test combine serial three counting and Timed up-and-go test simultaneously. It evaluates dual task performance.

SECONDARY OUTCOMES:
Change score of Depression, Anxiety Stress Scales-21 (DASS-21) | Baseline, immediate after treatment, 4-week follow up
  DASS-21 is a self-report questionnaire that measure symptoms of depression, anxiety, and stress.
Change score of Pittsburg Sleep Quality Index | Baseline, immediate after treatment, 4-week follow up
  PSQI is a self-report assessment which contains 19 items to measure sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chyi-Rong, Master, Principal Investigator — Chang gung memorial hospital, Kaohsiung branch
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung Medical Center, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No